CLINICAL TRIAL: NCT04900584
Title: A Prospective Randomized Multicenter Controlled Study to Optimize Heart Failure Care During TRANSitional Period in Patients With Acute Heart Failure With Reduced Ejection Fraction.
Brief Title: Optimize Heart Failure Care During TRANSitional Period in Patients With Acute Heart Failure.
Acronym: TRANS-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019ER630301
Record Dates: First submitted 2020-08-13; First posted 2021-05-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Acute Heart Failure
Keywords: Acute Heart Failure
MeSH Terms: interventions — Checklist; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group is managed by applying all three types of intervention.
  Interventions: Other: Checklist; Other: Education; Other: Telephone monitoring
- non-Intervention group (No Intervention): Non-intervention group is managed by conventional heart failure treatment.

INTERVENTIONS:
Other: Checklist — Checklist of guideline-based treatment before discharge
  Arms: Intervention group
Other: Education — Heart failure education before discharge
  Arms: Intervention group
Other: Telephone monitoring — Telephone monitoring after discharge
  Arms: Intervention group

SUMMARY:
The period of about a month after the discharge of acute heart failure patients is defined as a transition time. During this period, the patient has a high mortality rate and a readmission rate because the patient is not stabilized. In the United States and Europe, the readmission rate is more than 25% within 30 days, and the mortality rate within 30 days after discharge is three times that of patients with chronic heart failure.

The TRANS-HF is a prospective, randomized, multi-center, controlled study, which enrolls patients with acute heart failure with reduced ejection fraction.

The objective of TRANS-HF is to improve GAI at six months through three interventions: pre-discharge checklist, heart failure education, and telephone monitoring before the first outpatient visit.

ELIGIBILITY:
All consecutive hospitalized adult heart failure patients who fulfill one of 1-3 and satisfy 4-5 simultaneous

Inclusion Criteria:

1. Symptoms of heart failure
2. Signs of heart failure
3. Lung congestion in Chest-X-ray
4. Objective finding of structural and/or functional disorder of the heart or elevated natriuretic peptide levels
5. Left ventricular ejection fraction less than 40%

Exclusion Criteria:

1. Patients younger than 19 years old
2. Patients who do no consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Guideline adherence indicator at 6months | 6months
  the point of Guideline adherence indicator. Definition of GAI strata : Level of guideline-adherent treatment will be measured by guideline adherence indicator (GAI) such as 0/3, 1/3, 2/3, and 3/3. This GAI data will be obtained once after all prescription data has been collected. It will include whether or not prescribed medication of ≥50% of target dose : 0 points for non-prescription in the absence of contra-indications, 0.5 points for use of <50% of target dosage (<100% of target dose for MRA as the majority of patients were treated with ≥50% of target dose of MRA) or 1 point for use in ≥50% of target dosage (target dose for MRA). Non-administration of recommended drugs due to specific contraindications or intolerance will be scored as adherence to guidelines.

SECONDARY OUTCOMES:
Guideline adherence indicator at discharge | 0 day (at discharge)
  the point of Guideline adherence indicator. Definition of GAI strata : Level of guideline-adherent treatment will be measured by guideline adherence indicator (GAI) such as 0/3, 1/3, 2/3, and 3/3. This GAI data will be obtained once after all prescription data has been collected. It will include whether or not prescribed medication of ≥50% of target dose : 0 points for non-prescription in the absence of contra-indications, 0.5 points for use of <50% of target dosage (<100% of target dose for MRA as the majority of patients were treated with ≥50% of target dose of MRA) or 1 point for use in ≥50% of target dosage (target dose for MRA). Non-administration of recommended drugs due to specific contraindications or intolerance will be scored as adherence to guidelines.
Guideline adherence indicator at 1month | 1month after discharge
  the point of Guideline adherence indicator. Definition of GAI strata : Level of guideline-adherent treatment will be measured by guideline adherence indicator (GAI) such as 0/3, 1/3, 2/3, and 3/3. This GAI data will be obtained once after all prescription data has been collected. It will include whether or not prescribed medication of ≥50% of target dose : 0 points for non-prescription in the absence of contra-indications, 0.5 points for use of <50% of target dosage (<100% of target dose for MRA as the majority of patients were treated with ≥50% of target dose of MRA) or 1 point for use in ≥50% of target dosage (target dose for MRA). Non-administration of recommended drugs due to specific contraindications or intolerance will be scored as adherence to guidelines.
KCCQ(The Kansas City Cardiomyopathy Questionnaire) at discharge | 0 day (at discharge)
  the score of the Kansas City Cardiomyopathy Questionnaire
KCCQ(The Kansas City Cardiomyopathy Questionnaire) at 6 months | 6 months after discharge
  the score of the Kansas City Cardiomyopathy Questionnaire
EQ-5D(The EuroQoL five-dimensional instrument) at discharge | 0 day (at discharge)
  the score of the EuroQoL five-dimensional instrument
EQ-5D(The EuroQoL five-dimensional instrument) at 6 months | 6 months after discharge
  the score of The EuroQoL five-dimensional instrument
All-cause death | up to 6 months
  incidence rate (%) of death from any cause
Heart failure rehospitalization | up to 6 months
  incidence rate (%) of the first rehospitalization due to heart failure
Cardiovascular death | up to 6 months
  incidence rate (%) of death due to heart failure, arrhythmia and cerebrovascular event.
Cardiovascular rehospitalization | up to 6 months
  incidence rate (%) of the first rehospitalization due to heart failure, arrhythmia, and cerebrovascular event.
Composite end-point | up to 6 months
  incidence rate (%) of all-cause death and the first rehospitalization rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Su Yoo, MD, PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital,, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No